CLINICAL TRIAL: NCT02499133
Title: Identification and Comprehension of Focused Stress in a Sentence Among Adults Who Suffered Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-14-1031-HW-CTIL
Record Dates: First submitted 2015-01-08; First posted 2015-07-15 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-07

CONDITIONS: Focused Stress
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- adult who suffered traumatic brain injury (Other)
  Interventions: Other: language and cognitive tests
- control group (Other)
  Interventions: Other: language and cognitive tests

INTERVENTIONS:
Other: language and cognitive tests — The participants will undergo seven different. The tests will include different cognitive and language examinations. The main test of the study will be The Hebrew Focused Stress Test (HFST). The HFST includes three subtests. The first subtest requires identification of the stressed word in a sentence based on psychoacoustic abilities alone. The second and the third subtests require understanding the meaning of focused stress in different contexts - lexical grammatical and pragmatic/social. The test includes forty eight recorded sentences. In each sentence one word is stressed. The participants will be asked to listen to the recordings and answer a closed question regarding the stressed word.

SUMMARY:
Researches that focus on the perception of prosodic elements among adult who suffered traumatic brain injury (TBI), focus on their ability to decipher intonation in order to understand an additional meaning of a sentence. According to these researches, adults who suffer from TBI, with no signs of Aphasia, have difficulty perceiving and deciphering intonation (Marquardt et al., 2001; Angeleri et al., 2008). The current research asks to broaden the knowledge in this domain by examining the ability of adults with TBI to understand an additional prosodic element - focused stress.

The ability to identify and understand focused stress in a sentence requires different abilities. First, a psychoacoustic ability in order to detect the stressed word. Second, an ability to understand the lexical grammatical meaning of the word as it negates other possible meanings (for example, in the sentence "I'm eating a red apple" the stressed word negated the option of a different color). Third, an understanding of the stressed word as it creates a different pragmatic/social meaning (for example, in the sentence "mom, I asked for red, yellow and green candy" the role of the stressed word is to mark the candy that the addressee didn't get).

The aim of the study is to assess the ability of adults who had experienced TBI to grasp and understand the meaning of focused stress in the different contexts that were described above. An additional aim is to examine if differences in speech and cognitive abilities can describe some of the variation in the results.

Thirty adults between the ages of 18-50 years will take part in this study, fifteen adults who had experienced moderate to severe TBI (0.5-3 years post injury) and fifteen healthy adults. Each participant with TBI will be matched to a healthy adult by gender, age, education and social-economic status. All of the participants will be Hebrew native speakers, with no learning disability, no neurological injury, proper speech abilities and no hearing impairment.

The participants will undergo seven different tests in three different meetings (60 minute each), in a quiet room at Sheba - Academic Medical Center Hospital. The tests will include different cognitive and language examinations. The main test of the study will be The Hebrew Focused Stress Test (HFST). The HFST includes three subtests. The first subtest requires identification of the stressed word in a sentence based on psychoacoustic abilities alone. The second and the third subtests require understanding the meaning of focused stress in different contexts - lexical grammatical and pragmatic/social. The test includes forty eight recorded sentences. In each sentence one word is stressed. The participants will be asked to listen to the recordings and answer a closed question regarding the stressed word.

ELIGIBILITY:
Inclusion Criteria:

* Severity between moderate - severe as measured by the Glascow Coma Scale and time of PTA.
* Hebrew native speakers.
* between the ages of 18-50 years old.
* with no history of head trauma.
* with no history of use of addictive substance.
* with no history of psychiatric disorder.
* with no history of language disorder or language learning disability.
* with no degenerative cognition.
* are not suffering from aphasia.
* with a vision good enough to perform the tests of the study.
* with no hearing impairment.
* with a reading ability that is good enough to perform the test of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The Hebrew Focused Stress Test (HFST) | 15 min
  The HFST includes three subtests. The first subtest requires identification of the stressed word in a sentence based on psychoacoustic abilities alone. The second and the third subtests require understanding the meaning of focused stress in different contexts - lexical grammatical and pragmatic/social. The test includes forty eight recorded sentences. In each sentence one word is stressed. The participants will be asked to listen to the recordings and answer a closed question regarding the stressed word.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel